CLINICAL TRIAL: NCT00828958
Title: Local Site Tolerability of Multiple Dose Treatment With Deltoid Intramuscular Injection of RISPERDAL CONSTA in Subjects With Chronic Schizophrenia.
Brief Title: Injection Site Tolerability of Multiple Dose Treatment With Long-acting Injectable Risperidone Administered Via Deltoid Muscle in Chronic Schizophrenia Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011533
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Risperidone; Long acting injectable; Intradeltoidal injection
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Risperidone long-acting injectable

SUMMARY:
The purpose of this study is to examine the discontinuation rate of schizophrenia patients receiving multiple sequential 2 mL injections of long acting injectable risperidone (an atypical antipsychotic medication) when administered into the deltoid muscle once every 2 weeks.

DETAILED DESCRIPTION:
This is an open-label, multiple-dose, multicenter study in chronic schizophrenia patients, who are receiving long-acting injectable risperidone 25 or 37.5-mg injections into the gluteal muscle, and clinically require a higher dose. The study consists of a pretreatment screening phase, an 8-week, open label treatment phase during which patients will receive 4 sequential 2 mL injections with long-acting injectable risperidone (37.5 or 50 mg) administered every 2 weeks into the deltoid muscle in alternate arms (right versus left) for each visit; and a post treatment phase consisting of end of study evaluations upon completion of all the study procedures on Day 57 or at early withdrawal. The study hypothesis is that repeated injections of long-acting injectable risperidone into the deltoid muscle will be safe and well tolerated as assessed by the percent of patients who discontinue after at least 2 injections. Safety was assessed using adverse events (including occurrence of extrapyramidal symptoms as assessed by the Extrapyramidal Symptoms Rating Scale), clinical laboratory tests (hematology, serum chemistry, urinalysis, and pregnancy testing), vital signs, physical examinations, electrocardiograms, and injection site evaluation. The patients will receive 4 injections with long-acting injectable risperidone (37.5 or 50 mg) administered as 1 injection every 2 weeks into the deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

* Chronic schizophrenia of any subtype, according to DSM-IV criteria
* under current treatment with long-acting injectable risperidone 25 mg or 37.5 mg gluteal injections in an adequate study for at least 2 injections, and in need of a dose increase of long-acting injectable risperidone for clinical reason
* informed consent signed by the patient
* patient is otherwise healthy on the basis of a prestudy physical examination and medical history.

Exclusion Criteria:

* No DSM IV Axis I diagnosis other than schizophrenia
* no pregnant or breast feeding women
* no female subject of childbearing potential without adequate contraception
* no history of severe drug allergy or hypersensitivity
* no patients with inadequate mass in the deltoid regions to receive the intramuscular drug injections.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who discontinued from the study after having received at least 2 deltoid injections will be recorded.

SECONDARY OUTCOMES:
Reasons for discontinuation, patient rated local site injection pain and investigator rated local site injection reaction will be assessed at predefined times throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Injection site tolerability of multiple dose treatment with long-acting injectable risperidone administered via deltoid muscle in chronic schizophrenia patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=735&filename=CR011533_CSR.pdf